CLINICAL TRIAL: NCT04858763
Title: The Impact of the COVID-19 Pandemic on the Reporting and Management of Multiple Sclerosis Relapses
Brief Title: MS Relapses During COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 21NS011
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Multiple Sclerosis; Covid19; Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; COVID-19; Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2020 Cohort: This is the 2020 MS cohort who experienced a clinician confirmed relapse during April - June 2020, during the first wave of the COVID-19 pandemic.
  Interventions: Other: No Intervention
- 2019 Cohort: 2019 MS cohort who experienced a clinician confirmed relapse during April - June 2019.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — There will be no intervention during this study.

SUMMARY:
Throughout the COVID-19 pandemic, and to our knowledge there have been no studies looking systematically at the occurrence of MS relapses and their subsequent management, during the peak of the first wave of the pandemic. In this study we will explore how MS relapses were reported and managed during April - June 2020, compared to a control cohort who experienced a relapse during the same period in 2019 across 5 UK centers.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic inflammatory, demyelinating and neurodegenerative condition of the central nervous system (CNS) and is considered the most common cause of disability in young adults. It is estimated that the number of adults with MS in the UK has risen to 131,720. The majority of patients (85%) have Relapsing Remitting MS (RRMS), with many later entering the secondary progressive phase (SPMS). Relapse is the cardinal clinical feature of RRMS, and can be also prevalent in SPMS, however the influence of relapses on the long-term disability is not yet fully defined and remains controversial.

Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) emerged in Wuhan, China, in late 2019 and Covid-19, a disease caused by SARS-CoV-2 became a pandemic in March 2020. The impact of SARS-CoV-2 infection on patients with MS has yet to be elucidated. The main focus of previous studies has been the actual risk of Covid-19 inpatients with MS, the risk of MS exacerbation during Covid-19 infection and the impact of disease modifying drugs (DMDs) in the severity of Covid-19 infection. Other studies have explored the psychological and behavioural impact of Covid-19 pandemic to MS patients; those studies highlighted the risks from missing/cancelling clinic appointments and MRIs, missing/stopping/changing DMDs, delays in DMDs infusions, having a relapse and not seeking medical advice or disruptions in rehabilitation services. To the best of our knowledge, there is currently no study that explored the effect of Covid-19 on MS patients by looking systematically into MS relapses and their potential consequences. We will study the occurrence and subsequent management of relapses occurring between April - June 2020 at the peak of the first wave of the pandemic, compared to individuals who have relapsed during the same period in 2019. This observational, retrospective study will be performed at 5 UK sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of MS or Clinically Isolated Syndrome (CIS) and
* Atleast one clinician confirmed probable relapse between 01/04/2020 and 30/06/2020 or 01/04/2019 and 30/06/2019

Exclusion Criteria:

* Age <16 years

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All individuals with MS or CIS being treated by the respective UK sites will be screened for inclusion in this study.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Compare the number of MS relapses during the first wave of the Covid-19 pandemic to the same period in 2019. | 01/04/2020 and 30/06/2020 or 01/04/2019 and 30/06/2019

SECONDARY OUTCOMES:
1. To compare decisions made about administration of DMDs (starting or switching to a DMD) when a patient with MS has a relapse during the Covid-19 pandemic and in the same period in 2019. | 01/04/2020 and 30/06/2020 or 01/04/2019 and 30/06/2019
2. To compare decisions around treating an MS relapse with steroids during the Covid-19 pandemic and the same period in 2019. | 01/04/2020 and 30/06/2020 or 01/04/2019 and 30/06/2019

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Evangelou, Principal Investigator — University of Nottingham

IPD SHARING:
Plan to Share IPD: No
There is no plan to share any identifiable patient data.